CLINICAL TRIAL: NCT00990938
Title: A Phase 1, Multi-center, Randomized, Double-Blind, Placebo-controlled, Dose-escalation Safety Assessment Study of Combination Treatment With IMO-2125 and Ribavirin in Naïve Hepatitis C-infected, Genotype 1 Patients
Brief Title: Study of Combination Treatment With IMO-2125 and Ribavirin in Naïve Hepatitis C-infected, Genotype 1 Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMO-2125-201
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Hepatitis C, Treatment Naïve, Genotype 1 Patients
MeSH Terms: conditions — Hepatitis C | interventions — tilsotolimod; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): If randomized to placebo the patient will receive a subcutaneous injection once per week for 4 weeks
  Interventions: Drug: Saline
- IMO-2125 (Experimental): If randomized to receive the experimental treatment, IMO-2125, the patient will receive a subcutaneous injection once per week for 4 weeks
  Interventions: Drug: IMO-2125

INTERVENTIONS:
Drug: IMO-2125 — IMO 2125 is a synthetic DNA-based agonist of Toll-like receptor 9, which is expressed in humans in plasmacytoid dendritic cells and B cells of the immune system.
  Arms: IMO-2125
Drug: Saline — Subcutaneous injection once per week for four weeks
  Arms: Saline

SUMMARY:
Phase 1, randomized, double-blind, placebo-controlled, dose-escalation study with 3 dose levels of IMO-2125 in combination with standard weight based ribavirin (investigational treatment arm) or placebo in combination with ribavirin (RBV). Each cohort of 15 patients will be randomized 4:1 to receive the investigational treatment arm (12 patients) or placebo and RBV arm (3 patients).

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled, dose-escalation study with 3 dose levels of IMO-2125 in combination with standard ribavirin or placebo plus ribavirin. Each cohort will be randomized 4:1 to receive the investigational treatment arm or placebo and ribavirin. Three varying dose levels of IMO-2125 will be included. In both arms, ribavirin will be dosed based on patient weight.

Approximately 50 patients will be enrolled in France and Russia. Patients will provide informed consent prior to any screening procedures being performed. Screening will occur within 21 days prior to randomization. Enrolled patients who qualify and proceed successfully through the screening period will be randomized to receive 4 weeks of either the investigational treatment arm (IMO-2125 and ribavirin) or placebo and ribavirin, with a 4 week follow-up period.

Patients who are randomized to the investigational treatment arm will receive one of 3 dose levels of IMO 2125 SC once weekly; each patient will receive the same dose throughout the 4 weeks of treatment. In addition to IMO-2125 treatment they will also receive daily ribavirin, which will be given based on the patients weight and will be taken twice daily for a total of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented genotype 1
* HCV-positive with documented detectable plasma viral concentration > 10,000 IU/mL

Exclusion Criteria:

* Positive test for HIV or HbsAg
* Inadequate bone marrow, liver, and renal function
* Treatment with any IFN-based or other experimental or antiviral therapies - prior or current
* Other significant medical disease
* Concurrent or planned treatment during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Ribavirin: Placebo cohort: Saline (placebo) sc once weekly + Ribavirin (1000 mg dose for patients <75 kg; 1200 mg dose for patients ≥75 kg) administered orally in 2 divided oral doses.
- IMO-2125 0.08 mg/kg Weekly + Ribavirin: First experimental cohort: IMO-2125 0.08 mg/kg weekly + Ribavirin (1000 mg dose for patients <75 kg; 1200 mg dose for patients ≥75 kg), administered orally in 2 divided oral doses.
- IMO-2125 0.16 mg/kg Weekly + Ribavirin: Second experimental cohort: IMO-2125 0.16 mg/kg weekly + Ribavirin (1000 mg dose for patients <75 kg; 1200 mg dose for patients ≥75 kg), administered orally in 2 divided oral doses.
- IMO-2125 0.32 mg/kg Weekly + Ribavirin: Third experimental cohort: IMO-2125 0.32 mg/kg weekly + Ribavirin (1000 mg dose for patients <75 kg; 1200 mg dose for patients ≥75 kg), administered orally in 2 divided oral doses.
- IMO-2125 0.16 mg/kg Twice Weekly + Ribavirin: Fourth experimental cohort: IMO-2125 0.16 mg/kg twice weekly + Ribavirin (1000 mg dose for patients <75 kg; 1200 mg dose for patients ≥75 kg), administered orally in 2 divided oral doses.
- Peg-rIFN + Ribavirin: Active comparator cohort: Peg-rIFN 180 µg sc once weekly + Ribavirin (1000 mg dose for patients <75 kg; 1200 mg dose for patients ≥75 kg) administered orally in 2 divided oral doses.
Period: Overall Study
Arm/Group | Placebo + Ribavirin | IMO-2125 0.08 mg/kg Weekly + Ribavirin | IMO-2125 0.16 mg/kg Weekly + Ribavirin | IMO-2125 0.32 mg/kg Weekly + Ribavirin | IMO-2125 0.16 mg/kg Twice Weekly + Ribavirin | Peg-rIFN + Ribavirin
Started | 3 | 12 | 12 | 12 | 12 | 12
Completed | 3 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Ribavirin | IMO-2125 0.08 mg/kg Weekly + Ribavirin | IMO-2125 0.16 mg/kg Weekly + Ribavirin | IMO-2125 0.32 mg/kg Weekly + Ribavirin | IMO-2125 0.16 mg/kg Twice Weekly + Ribavirin | Peg-rIFN + Ribavirin | Total
Number analyzed (Participants) | 3 | 12 | 12 | 12 | 12 | 12 | 63
Age, Continuous [Median (Full Range); unit: years] | 30.0 [28 to 52] | 40.5 [28 to 57] | 38.0 [19 to 47] | 48.5 [23 to 57] | 42.5 [32 to 65] | 32.0 [26 to 64] | 39.0 [19 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 5 | 7 | 3 | 24
  Male | 1 | 9 | 8 | 7 | 5 | 9 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 12 | 11 | 12 | 12 | 12 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 22.4 [19.7 to 25.4] | 24.3 [20.5 to 32.7] | 22.7 [18.1 to 27.5] | 27.3 [22.8 to 38.7] | 24.1 [20.3 to 30.9] | 24.9 [21.7 to 31.1] | 24.8 [18.1 to 38.7]

OUTCOME MEASURES:

1. Primary Outcome: At Least 1 TEAE
Description: The number and percentage of subjects who experienced at least one treatment-emergent adverse event by category.
Time Frame: From first dose of study treatment to day 59 (end of study)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Ribavirin | IMO-2125 0.08 mg/kg Weekly + Ribavirin | IMO-2125 0.16 mg/kg Weekly + Ribavirin | IMO-2125 0.32 mg/kg Weekly + Ribavirin | IMO-2125 0.16 mg/kg Twice Weekly + Ribavirin | Peg-rIFN + Ribavirin
Number analyzed (Participants) | 3 | 12 | 12 | 12 | 12 | 12
Participants
  At least 1 TEAE | 2 | 12 | 12 | 12 | 12 | 12
  At least 2 TEAE related to study drug | 2 | 12 | 12 | 12 | 12 | 12
  At least 1 severe/life threatening TEAE | 0 | 2 | 7 | 2 | 3 | 7
  At least 1 injection site reaction | 0 | 12 | 12 | 11 | 12 | 9
  At least 1 TEAE that led to discontinuation | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment to day 59 (end of study)
Arm/Group | Placebo + Ribavirin | IMO-2125 0.08 mg/kg Weekly + Ribavirin | IMO-2125 0.16 mg/kg Weekly + Ribavirin | IMO-2125 0.32 mg/kg Weekly + Ribavirin | IMO-2125 0.16 mg/kg Twice Weekly + Ribavirin | Peg-rIFN + Ribavirin
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/12 | 7/12 | 2/12 | 3/12 | 11/12
Other Adverse Events (participants affected / at risk) | 2/3 | 12/12 | 12/12 | 12/12 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Ribavirin (N=3) | IMO-2125 0.08 mg/kg Weekly + Ribavirin (N=12) | IMO-2125 0.16 mg/kg Weekly + Ribavirin (N=12) | IMO-2125 0.32 mg/kg Weekly + Ribavirin (N=12) | IMO-2125 0.16 mg/kg Twice Weekly + Ribavirin (N=12) | Peg-rIFN + Ribavirin (N=12)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 6
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flu like symptoms (General disorders) | 0 | 0 | 2 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Ribavirin (N=3) | IMO-2125 0.08 mg/kg Weekly + Ribavirin (N=12) | IMO-2125 0.16 mg/kg Weekly + Ribavirin (N=12) | IMO-2125 0.32 mg/kg Weekly + Ribavirin (N=12) | IMO-2125 0.16 mg/kg Twice Weekly + Ribavirin (N=12) | Peg-rIFN + Ribavirin (N=12)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 1 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 7 | 2 | 7 | 10
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 0 | 8 | 10
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 4 | 4 | 5 | 3
Chills (General disorders) | 1 | 5 | 0 | 3 | 4 | 1
Fatigue (General disorders) | 1 | 3 | 1 | 1 | 1 | 0
Influenza-like illness (General disorders) | 1 | 5 | 8 | 3 | 5 | 8
Injection site discoloration (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 12 | 11 | 12 | 9
Injection site hematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Injection site induration (General disorders) | 0 | 0 | 7 | 8 | 9 | 3
Injection site pain (General disorders) | 0 | 0 | 11 | 9 | 10 | 3
Injection site pruritus (General disorders) | 0 | 1 | 3 | 3 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 8 | 4 | 11 | 9 | 5
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 4 | 7 | 4 | 2 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0
Urobilin urine present (Investigations) | 0 | 2 | 1 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 3 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 3 | 4 | 2
Headache (Nervous system disorders) | 1 | 8 | 1 | 2 | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Purritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes